CLINICAL TRIAL: NCT07142980
Title: A Phase I Study of HRS-7172 Evaluating Safety, Tolerability and Pharmacokinetics in Participants With Advanced Solid Tumors Harboring RAS Mutations or Amplifications
Brief Title: A Phase I Study of HRS-7172 in Participants With Advanced Solid Tumors Harboring RAS Mutations or Amplifications
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7172-101
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors Harboring RAS Mutations or Amplifications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-7172 Group (Experimental): Oral HRS-7172.
  Interventions: Drug: HRS-7172 Tablets

INTERVENTIONS:
Drug: HRS-7172 Tablets — HRS-7172 tablets.

SUMMARY:
This is a phase I study of HRS-7172 to evaluate safety, tolerability and pharmacokinetics in participants with advanced solid tumors harboring RAS mutations or amplifications.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood this study and are willing to sign the ICF, with good compliance and cooperation in follow-up;
2. Aged between 18-75 years old;
3. ECOG performance status (PS) score of 0 or 1;
4. Life expectancy > 3 months;
5. At least one measurable lesion per RECIST v1.1;
6. Adequate organ function.

Exclusion Criteria:

1. Toxicity from prior anti-tumor treatment has not recovered to Grade ≤ 1 or a level specified in the inclusion/exclusion criteria;
2. Presence of central nervous system (CNS) metastases;
3. Participants with gastrointestinal diseases that affect drug administration/absorption;
4. Participants who have undergone major surgery other than diagnosis or biopsy within 28 days before the first dose, or are expected to undergo major surgery during the study period;
5. Presence of serious pulmonary diseases;
6. Active tuberculosis or a history of active tuberculosis infection within 48 weeks prior to screening, regardless of whether they have been treated;
7. Active or persistent gastrointestinal bleeding within 6 months prior to screening;
8. History of allogeneic bone marrow or solid organ transplantation;
9. History of deep vein thrombosis or pulmonary embolism within 6 months prior to screening;
10. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring clinical intervention;
11. Positive human immunodeficiency virus (HIV) (HIV1/2 antibodies), active chronic hepatitis B, or active hepatitis C (positive HCV antibody and positive HCV RNA);
12. Known history of hypersensitivity to any component of the drug product to be used in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From screening period up to 30 days after the last dose.
Incidence and severity of serious adverse events (SAEs) | From screening period up to 30 days after the last dose.
Dose-limiting toxicity (DLT) | From day 1 to day 24.
Maximum tolerated dose (MTD) | From day 1 to day 24.
Recommended Phase II Dose (RP2D) | From day 1 to day 24.

SECONDARY OUTCOMES:
Objective response rate (ORR) | About 24 months.
Duration of response (DoR) | About 24 months.
Disease control rate (DCR) | About 24 months.
Progression-free survival (PFS) | About 24 months.
Overall survival (OS) | About 24 months.
Maximum plasma concentration (Cmax) | About 24 months.
Time to maximum concentration (Tmax) | About 24 months.
Elimination half-life (t1/2) | About 24 months.
Area under concentration-time curve from time 0 to the last measurable concentration time point t (AUC0-t) | About 24 months.
Area under concentration-time curve from time 0 to infinity (AUC0-∞) | About 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Affiliated Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided